CLINICAL TRIAL: NCT03707561
Title: Russian National Registry of Patients With Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension
Brief Title: RUS-registry of PH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Russian Cardiology Research and Production Center (Other)
Collaborators: Scientific Research Institute of Rheumatology (Unknown)
Responsible Party: Principal Investigator, Tamila V. Martynyuk, MD, PhD, Russian Cardiology Research and Production Center, Russian Cardiology Research and Production Center
Other Study IDs: NMIC for Cardiology
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Group 1 - IPAH and heritable PAH: Idiopathic pulmonary arterial hypertension (IPAH) and heritable PAH Diagnostic Test: Right Heart Catheterization (RHC)
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC)
- Group 2- PAH associated with CHD: Pulmonary arterial hypertension associated with congenital heart disease Diagnostic Test: Right Heart Catheterization (RHC)
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC)
- Group 3- PAH associated with CTD: Pulmonary Arterial Hypertension associated with Connective Tissue Diseases Diagnostic Test: Right Heart Catheterization (RHC)
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC)
- Group 4- portoPH: Portopulmonary hypertension
- group 5- PAH-HIV: Pulmonary arterial hypertension associated with HIV infection
- group 6- operable CTEPH: Operable chronic thromboembolic pulmonary hypertension Diagnostic Test: Right Heart Catheterization (RHC)
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC)
- group 7- non-operable CTEPH: Non operable chronic thromboembolic pulmonary hypertension Diagnostic Test: Right Heart Catheterization (RHC)
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC)

INTERVENTIONS:
Diagnostic Test: Right Heart Catheterization (RHC) — RHC at the enrollment and every 12 months
  Groups: Group 1 - IPAH and heritable PAH; Group 2- PAH associated with CHD; Group 3- PAH associated with CTD; group 6- operable CTEPH; group 7- non-operable CTEPH

SUMMARY:
Russian National Registry of Patients With Pulmonary Arterial Hypertension (PAH) and Chronic Thromboembolic Pulmonary Hypertension (CTEPH) is a multicenter, observational study of the clinical course and disease management of PAH and CTEPH patients. designed to gather demographic, clinical and prognostic data of routine medical care in prospective manner for newly initiated treatment since Jan 2016.

The internet-based registry (www.medibase.pro) fulfills high quality standards through several measures (planned minimum centre contribution of at least 10 patients per year, automated plausibility checks of data at entry, queries, monitoring with source data verification in >50% of participating centers).

All consecutive patients diagnosed with World Health Organization Pulmonary Hypertension Groups (WHO Group I) PAH according to specific hemodynamic criteria will be enrolled in participating centers after signing the informed consents. Participating patients will be followed for a minimum of five years from the time of enrollment.

It can be applied, among further purposes, for quality assurance: individual centers can confidentially compare their results with the combined outcome of the other centers. It is expected that the registry contributes to optimization of specific drug therapy for PAH and Pulmonary Hypertension (PH).

DETAILED DESCRIPTION:
Russian National Registry of Patients With Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension (RUS-registry of PH) will report current and comprehensive data on

* Demographics, clinical course of incident PAH and CTEPH, the hemodynamic and functional status of patients
* The main diagnostic approaches for the diagnosis of PAH and CTEPH.
* Patient outcomes including survival, by subgroup, by treatment strategy and other factors
* Clinical predictors of short-term and long-term clinical outcomes
* Relationship between PAH- treatment medications and patient outcomes
* Temporal trends in treatments and outcomes for newly diagnosed patients
* The state of implementation of current PAH guidelines
* To describe the status of operable or non-operable patients with PAH and CTEPH
* To identify the most important prognostic indicators in patients with PH.
* To study the basic principles of therapy of patients with PH.patients
* To evolve research needs of the PAH community

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed PAH:

idiopathic form (IPAH) or PAH associated with connective tissue diseases (PAH-CTD), with congenital heart defects (PAH-CHD), with HIV infection (PAH-HIV), or portopulmonary hypertension Newly diagnosed CTEPH- operable and non-operable

Documentation of the following hemodynamic parameters by right heart catheterization, performed at the time of study enrollment:

Mean pulmonary arterial pressure (mPAP) ≥ 25 mm Hg at rest Pulmonary wedge pressure < 15 mm Hg Pulmonary vascular resistance (PVR) ≥ 240 dynes.sec.cm-5 (i.e., ≥ 3.0 Wood units) Signed informed consent Previously naïve patients with newly initiated therapy with endothelin receptor antagonists (ERA), phoshodiesterase-5 (PDE-5) inhibitors, soluble guanylate cyclase (sGC) stimulators or prostacyclins in mono- or combination therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IPAH and heritable PAH, PAH associated with CHD, PAH associated with CTD, portoPH, PAH-HIV, operable CTEPH, non-operable CTEPH
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
RHC | 12 month
  Change of pulmonary vascular resistance

CONTACTS AND LOCATIONS:
Overall Officials: Tamila Martynyuk, MD, PhD, Principal Investigator — Russian Cardiology Research and Production Center; Irina Chazova, MD, PhD, Study Chair — Russian Cardiology Research and Production Center; Olga Arkhipova, PhD, Study Director — Russian Cardiology Research and Production Center; Alexander Volkov, MD, PhD., Study Director — Institute of Rheumatology named after VA Nasonova, Moscow, Russia; Vera Lukyantchikova, MD, PhD, Study Director — Regional Clinical Hospital №1, Khabarovsk, Russia; Elena Vetrova, PhD, Study Director — Belgorod Regional Clinical Hospital, Belgorod, Russia; Elena Devitiyarova, MD, PhD, Study Director — Rostov Regional State CLINICAL HOSPITAL, Russia; Olga Korolkova, MD, PhD, Study Director — Department of Hospital Therapy of the Voronezh State Medical Academy. N. N. Burdenko, Voronezh, Russia; Olga Andreyeva, Study Director — State Healthcare Institution Regional Cardiology Dispensary, Ulyanovsk, Russia; Svetlana Martynenko, Study Director — Regional Budget Cardiology Dispensary, Astrakhan, Russia; Elena Milovanova, PhD, Study Director — District Cardiology Dispensary "Center for Diagnostic and Cardiovascular Surgery", Surgut, Russia; Anna Rogacheva, Study Director — State Future Health Care Institution "Primorskaya Regional Clinical Hospital № 1", Vladivostok, Russia; Svetlana Kharitonova, Study Director — State budgetary health care institution "Bryansk Regional Cardiology Dispensary", Bryansk, Russia; Elena Shutemova, MD, PhD, Study Director — IVANOVO STATE MEDICAL ACADEMY Department of Therapy and General Practice, Ivanovo, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chazova IE, Martynyuk TV. [Clinical guidelines for the diagnosis and treatment of chronic thromboembolic pulmonary hypertension (Part 1)]. Ter Arkh. 2016;88(9):90-101. doi: 10.17116/terarkh201688990-101. Russian. PMID 27735920
- [Background] Chazova IE, Martynyuk TV. [Clinical guidelines for the diagnosis and treatment of chronic thromboembolic pulmonary hypertension (Part 2)]. Ter Arkh. 2016;88(10):63-73. doi: 10.17116/terarkh201688663-73. Russian. PMID 27801422
- [Background] Chazova IE, Avdeev SN, Tsareva NA, Volkov AV, Martyniuk TV, Nakonechnikov SN. [Clinical guidelines for the diagnosis and treatment of pulmonary hypertension]. Ter Arkh. 2014;86(9):4-23. Russian. PMID 25518501
- [Result] Taran IN, Belevskaya AA, Saidova MA, Martynyuk TV, Chazova IE. Initial Riociguat Monotherapy and Transition from Sildenafil to Riociguat in Patients with Idiopathic Pulmonary Arterial Hypertension: Influence on Right Heart Remodeling and Right Ventricular-Pulmonary Arterial Coupling. Lung. 2018 Dec;196(6):745-753. doi: 10.1007/s00408-018-0160-4. Epub 2018 Sep 4. PMID 30182153
- [Result] Chazova IE, Arkhipova OA, Valieva ZS, Nakonechnikov SN, Martyniuk TV. [Pulmonary hypertension in Russia: the first results of the national register]. Ter Arkh. 2014;86(9):56-64. Russian. PMID 25518507
- See also: First date of Russian national registry of pulmonary arterial hypertension — https://doi.org/10.1097/01.hjh.0000467958.52984.9f